CLINICAL TRIAL: NCT02853734
Title: Comparative Evaluation of the Inflammatory Status of Visceral Adipose Tissue From Obese Patients According to the Presence and Severity of Periodontitis
Brief Title: Inflammatory Status of Visceral Adipose Tissue in Obese Patients Related to Periodontitis Severity
Acronym: BACTERIOB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2015/CHU/13
Record Dates: First submitted 2016-07-26; First posted 2016-08-03 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Parodontitis; Obesity; Metabolism Disorders
MeSH Terms: conditions — Dry Socket; Obesity; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEVERE PERIODONTITIS (Experimental): Periodontal examination Biological samples collection: periodontal, saliva, blood, fecal, visceral adipose tissue
  Interventions: Other: SEVERE PERIODONTITIS
- NO PERIODONTITIS (Other): Periodontal examination Biological samples collection: periodontal, saliva, blood, fecal, visceral adipose tissue
  Interventions: Other: NO PERIODONTITIS

INTERVENTIONS:
Other: SEVERE PERIODONTITIS — Patients exhibiting moderate to severe periodontitis
  Arms: SEVERE PERIODONTITIS
Other: NO PERIODONTITIS — Patients without existing periodontitis or exhibiting mild periodontitis
  Arms: NO PERIODONTITIS

SUMMARY:
The research aims to compare the inflammatory status of visceral adipose tissue from obese patients depending on the presence and severity of periodontitis, in order to establish a potential causal link between the severity of the bacterial contamination and insulin resistance.

DETAILED DESCRIPTION:
Recruitment of patients will be achieved in the department of digestive surgery. It will involve 122 patients with severe obesity undergoing bariatric surgery scheduled within the digestive surgery department. Patients recruited will be examined for evaluating the presence and severity of periodontitis, and separated into either group 1: for patients with moderate or severe periodontitis, and or group 2: for patients without or with mild periodontitis. The day before the surgery, blood sample will be collected for the analysis of circulating metabolic and inflammatory markers. Collection of stimulated saliva, periodontal sample and faeces samples (50 g) will also be carried out for bacteria determination. During the surgical procedure, a sample of visceral adipose tissue (50 g) will be collected and used for periodontal bacteria detection and inflammatory markers analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for bariatric surgery scheduled within the digestive surgery
* Patient affiliated to Social Security system or equivalent

Exclusion Criteria:

* Treatment with steroids or anti-inflammatory drugs in progress (or stopped for less than one month)
* Patients who received antibiotics within 3 months prior to the bariatric surgery for whatever duration
* Dental current (or older than 3 months)
* Participation in another research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Inflammatory status of visceral adipose tissue from obese patients depending on the presence and severity of periodontitis | Consecutively to visceral fat biopsy (day of surgery)
  Measurements of major adipocytokines (Interleukine 6, Leptin, Adiponectin, Tumor Necrosis Factor-alpha, Monocyte Chemoattractant Protein-1, macrophage F4/80 receptor, CD11c, nuclear factor-kappa B, Toll Like Receptor 2/4 )

SECONDARY OUTCOMES:
Detection of DNA for at least one type of periodontal pathogens in adipose tissue | Consecutively to visceral fat biopsy (day of surgery)
  Aggregatibacter actinomycetemcomitans, Fusibacterium nucleatum, Porphyromonas gingivalis, Prevotella intermedia, Treponema denticola and Tannerella forsythia
Description of the metabolic profile of patients relative to periodontitis severity | Consecutively to periodontal examination (day before surgery)
  glycemia, insulinemia, glucose tolerance, plasma and HDL total cholesterol, triglycerides
Link between adipose tissue inflammatory status, bacterial contamination and metabolic profile of patients | Consecutively to periodontal examination and fat biopsy (day before surgery, day of surgery)
  adipose tissue inflammatory status, periodontal bacterial contamination,diabetic disorders, lipid metabolic profile of patients
Link between the presence of periodontal pathogens in adipose tissue and their detection in saliva and plasma | Consecutively to periodontal examination and fat biopsy (day before surgery, day of surgery)
  Detection of antibodies directed to periodontal bacteria in saliva and plasma

OTHER OUTCOMES:
Collection of biological samples | Consecutively to samples collection (day before surgery, day of surgery)
  Plasma, saliva and adipose tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No